CLINICAL TRIAL: NCT00742001
Title: IMPROVE: Inactivation of Whole Blood With Mirasol (R): Performance in Red Blood Cells, Platelets and Plasma Investigation
Brief Title: Feasibility Study of Mirasol-Treated Whole Blood Red Cell Recovery and Survival
Acronym: IMPROVE
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: An endpoint difference between 3 energies was not observed at interim analysis
Sponsor: Terumo BCTbio (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CTS-0040
Record Dates: First submitted 2008-08-25; First posted 2008-08-27 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Healthy
Keywords: red blood cells; transfusion; recovery; feasibility; white blood cell inactivation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mirasol Illumination Dose #1 (Experimental): Whole blood units treated with Mirasol at Illumination dose #1 (A1) of 22 Joules per milliliter of red blood cells (J/mL RBCs)
  Interventions: Biological: Mirasol System for Whole Blood.
- Mirasol Illumination Dose #2 (Experimental): Whole Blood units treated with Mirasol at Illumination dose #2 (A2) of 33 J/mL RBCs
  Interventions: Biological: Mirasol System for Whole Blood.
- Mirasol Illumination Dose #3 (Experimental): Whole Blood units treated with Mirasol at Illumination dose #3 (A3) of 44 J/mL RBCs
  Interventions: Biological: Mirasol System for Whole Blood.

INTERVENTIONS:
Biological: Mirasol System for Whole Blood. — Treatment of whole blood with the Mirasol system at 3 experimental illumination energies for testing of autologous RBC recovery and survival in healthy subjects
  Other Names: Mirasol System; Mirasol

SUMMARY:
Feasibility trial to evaluate recovery and survival of red blood cells (RBCs) from Mirasol-treated whole blood

DETAILED DESCRIPTION:
Radiolabeling of red blood cells (RBCs) followed by infusion back to the donor is commonly used to test the quality of RBCs in a person. By measuring the level of radioisotope in a blood sample, these tests evaluate what percentage of the RBCs remain in the bloodstream after 24 hours (recovery) and can predict how long the RBCs will remain in circulation (survival). The IMPROVE trial is a feasibility trial to evaluate these parameters in RBCs obtained from whole blood units that have been treated with the Mirasol System.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults who meet AABB (formerly known as the American Association of Blood Banks) criteria for whole blood donation
* females incapable of becoming pregnant
* males agreeing to use contraception during trial

Exclusion Criteria:

* pregnancy or nursing
* abnormal medical history (bleeding disorders, anemia, myocardial ischemia, uncontrolled hypertension, heart disease, epilepsy)
* major surgery
* use of drugs affecting coagulation or RBC function
* recent participation in other trials which may confound results

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-09-10 (Actual); Primary Completion 2008-11-20 (Actual); Study Completion 2008-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Cancelas-Perez, M.D, Ph.D, Principal Investigator — University of Cincinnati, Hoxworth Blood Center
Locations (1):
- University of Cincinnati, Hoxworth Blood Center, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Mirasol Illumination Dose #1 (A1): Whole blood units treated with Mirasol at Illumination dose #1: 22 Joules per milliliter of red blood cells (J/mL RBC)
  Mirasol System for Whole Blood.: Treatment of whole blood with the Mirasol system at 3 experimental illumination energies for testing of autologous RBC recovery and survival in healthy subjects
- Mirasol Illumination Dose #2 (A2): Whole Blood units treated with Mirasol at Illumination dose #2: 33 J/mL RBC
  Mirasol System for Whole Blood.: Treatment of whole blood with the Mirasol system at 3 experimental illumination energies for testing of autologous RBC recovery and survival in healthy subjects
- Mirasol Illumination Dose #3 (A3): Whole Blood units treated with Mirasol at Illumination dose #3: 44 J/mL RBC
  Mirasol System for Whole Blood.: Treatment of whole blood with the Mirasol system at 3 experimental illumination energies for testing of autologous RBC recovery and survival in healthy subjects
Period: Overall Study
Arm/Group | Mirasol Illumination Dose #1 (A1) | Mirasol Illumination Dose #2 (A2) | Mirasol Illumination Dose #3 (A3)
Started | 4 | 4 | 4
Completed | 4 | 4 | 3
Not Completed | 0 | 0 | 1
Not completed — Withdrawn; health exclusion (flu) | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Mirasol Illumination Dose #1 (A1): Whole blood units treated with Mirasol at Illumination dose #1: 22 J/mL RBC
  Mirasol System for Whole Blood.: Treatment of whole blood with the Mirasol system at 3 experimental illumination energies for testing of autologous RBC recovery and survival in healthy subjects
- Total: Total of all reporting groups
Arm/Group | Mirasol Illumination Dose #1 (A1) | Mirasol Illumination Dose #2 (A2) | Mirasol Illumination Dose #3 (A3) | Total
Number analyzed (Participants) | 4 | 4 | 4 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 4 | 11
  >=65 years | 0 | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (7) | 42 (18) | 51 (13) | 46 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 5
  Male | 2 | 2 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 4 | 4 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 4 | 12
Height (inches) [Mean (Standard Deviation); unit: inches] | 69 (4) | 70 (3) | 68 (3) | 69 (3)
Weight (lbs) [Mean (Standard Deviation); unit: lbs] | 219 (26) | 180 (17) | 253 (62) | 217 (48)
Pulse (bpm) [Mean (Standard Deviation); unit: bpm] | 68 (5) | 68 (3) | 72 (11) | 69 (7)
Systolic Blood Pressure (mmHg) [Mean (Standard Deviation); unit: mmHg] | 123 (11) | 112 (11) | 122 (16) | 119 (13)
Diastolic Blood Pressure (mmHg) [Mean (Standard Deviation); unit: mmHg] | 76 (5) | 69 (7) | 76 (13) | 74 (9)
Oral Temperature degrees Fahrenheit (F) [Mean (Standard Deviation); unit: degrees Fahrenheit (F)] | 98 (0.6) | 97 (0.3) | 97 (0.4) | 97 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Red Blood Cell (RBC) Recovery
Description: The 24-hour recovery calculation was conducted to evaluate the percentage of labeled RBCs remaining in the circulation 24 hours after re-infusion of the cells, as compared to Time 0 measurements (time of re-infusion). FDA requires at least 75% recovery for new RBC processes.
Time Frame: 24-hour post autologous infusion of RBCs
Measure: Mean (Standard Deviation); unit: percentage of recovered RBCs
Arm/Group | Mirasol Illumination Dose #1 (A1) | Mirasol Illumination Dose #2 (A2) | Mirasol Illumination Dose #3 (A3)
Number analyzed (Participants) | 4 | 4 | 3
percentage of recovered RBCs | 77.8 (3.4) | 70.5 (7.5) | 68.1 (6.3)

2. Secondary Outcome: Predicted Total Lifespan of Red Blood Cells (RBCs), Based on 28-day RBC Survival
Description: The objective of measuring 28-day survival was to identify the potential total lifespan of labeled RBCs in circulation. Normal, native RBCs remain in circulation for a maximum of approximately 120 days; by using the 51Cr half-life of approximately 28 days, and its elution rate from labeled RBCs, the survival of the labeled cells can be predicted.
Time Frame: 28-days post autologous infusion of RBCs
Measure: Mean (Standard Deviation); unit: days
Groups:
- Mirasol Illumination Dose #1 (A1): Whole blood units treated with Mirasol at Illumination dose #1.
  Mirasol System for Whole Blood.: Treatment of whole blood with the Mirasol system at 3 experimental illumination energies for testing of autologous RBC recovery and survival in healthy subjects
- Mirasol Illumination Dose #2 (A2): Whole Blood units treated with Mirasol at Illumination dose #2.
  Mirasol System for Whole Blood.: Treatment of whole blood with the Mirasol system at 3 experimental illumination energies for testing of autologous RBC recovery and survival in healthy subjects
- Mirasol Illumination Dose #3 (A3): Whole Blood units treated with Mirasol at Illumination dose #3.
  Mirasol System for Whole Blood.: Treatment of whole blood with the Mirasol system at 3 experimental illumination energies for testing of autologous RBC recovery and survival in healthy subjects
Arm/Group | Mirasol Illumination Dose #1 (A1) | Mirasol Illumination Dose #2 (A2) | Mirasol Illumination Dose #3 (A3)
Number analyzed (Participants) | 4 | 4 | 3
days | 75.9 (17.8) | 66.9 (31.0) | 55.9 (20.6)

3. Secondary Outcome: Count of Participants With Serious Adverse Events (SAE)
Time Frame: 28-days post autologous infusion of RBCs
Measure: Count of Participants; unit: Participants
Arm/Group | Mirasol Illumination Dose #1 (A1) | Mirasol Illumination Dose #2 (A2) | Mirasol Illumination Dose #3 (A3)
Number analyzed (Participants) | 4 | 4 | 3
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the time of autologous RBC re-infusion until study completion (28 days)
Arm/Group | Mirasol Illumination Dose #1 (A1) | Mirasol Illumination Dose #2 (A2) | Mirasol Illumination Dose #3 (A3)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 1/4 | 2/4 | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirasol Illumination Dose #1 (A1) (N=4) | Mirasol Illumination Dose #2 (A2) (N=4) | Mirasol Illumination Dose #3 (A3) (N=4)
Slight heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Head stuffiness and congestion (allergy related) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cold, sore throat, sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus infection and bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Flu (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Two major limitations to the interpretation of these data. 1)the small sample size limited the interpretation of some of the data. 2)the high degree of inter-subject variability further limits the interpretation of potential trends seen in the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All publication of results and or design of this study are contingent upon approval from the sponsor.